CLINICAL TRIAL: NCT00481195
Title: An 8 Week Double Blind, Placebo-Controlled, Parallel Group, Fixed Dosage Study to Evaluate the Efficacy and Safety of Armodafinil Treatment (150mg/Day) as Adjunctive Therapy in Adults With Major Depression Associated With Bipolar I Disorder
Brief Title: Armodafinil Treatment as Adjunctive Therapy in Adults With Major Depression Associated With Bipolar I Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C10953/2032/DP/US; NCT00547222 (obsolete NCT alias)
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Results first posted 2010-12-20 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Bipolar I Depression
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Armodafinil (Active Comparator)
  Interventions: Drug: Armodafinil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Armodafinil — Patients were randomly assigned to begin oral treatment with armodafinil, which was titrated to 150 mg/day (3 tablets). Armodafinil was titrated up to the target dosage of 150 mg/day (daily dose was administered each morning). Patients began taking blinded armodafinil at a dose of 50 mg/day (1 tablet) on the day following the baseline visit. Doses were increased by 50 mg/day (1 tablet) to a dose of 100 mg/day on Day 2 and 3, and then again by 50 mg /day on day 4 for a target dose of 150 mg/day. Following titration, patients continued taking 150 mg/day of armodafinil for the duration of the study. If a patient was unable to tolerate (recurrent or persistent adverse events) the study drug, 1 reduction in dosage (ie, minimum dosage 100 mg/day [2 tablets]) was allowed. The dosage could not be increased after it was decreased.
  Arms: Armodafinil
Drug: Placebo — Patients were randomly assigned to begin oral treatment with placebo, which was titrated to 3 tablets. Placebo tablets matching the 50 mg armodafinil tablet were used in a manner identical to that of the armodafinil tablets. Study drug was titrated up to the target dosage of 3 tablets / day (daily dose was administered each morning). Patients began taking blinded study drug at a dose of 1 tablet daily on the day following the baseline visit. Doses were increased by 1 tablet to a dose of 2 tablets/day on Day 2 and 3, and then again by 1 tablet /day on day 4 for a target dose of 3 tablets/day. Following titration, patients continued taking 3 tablets/day of study drug for the duration of the study. If a patient was unable to tolerate (recurrent or persistent adverse events) the study drug, 1 reduction in dosage (ie, minimum dosage 2 tablets/day) was allowed. The dosage could not be increased after it was decreased.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine if armodafinil treatment, at a dosage of 150 mg/day, is more effective than placebo treatment as adjunctive therapy for adults who are experiencing a major depressive episode associated with Bipolar I Disorder and who are inadequately responsive to their current treatment for a current major depressive episode.

ELIGIBILITY:
Key Inclusion Criteria:

* The patient has a diagnosis of Bipolar I Disorder and is currently experiencing a major depressive episode.
* The patient is currently being treated with 1 or 2 of the following drugs: lithium, olanzapine, or valproic acid.

Key Exclusion Criteria:

* The patient has any Axis I disorder apart from Bipolar I Disorder that was the primary focus of treatment within 6 months before the screening visit (with the exception of nicotine dependence).
* The patient has any clinically significant uncontrolled medical or surgical condition.
* The patient has previously received modafinil or armodafinil, or the patient has a known sensitivity to any ingredients in the study drug tablets.
* The patient is a pregnant or lactating woman. (Any woman becoming pregnant during the study will be withdrawn from the study.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (42):
  - Birmingham Research Group, Birmingham, Alabama
  - Birmingham Psychiatry Pharmaceutical Studies, Inc, Birmingham, Alabama
  - Synergy Clinical Research Center, Escondido, California
  - Bay Area Research Institute, Lafayette, California
  - Synergy Clinical Research Center, National City, California
  - Excell Research, Oceanside, California
  - Pacific Clinical Research Medical Group, Orange, California
  - CNRI Los Angeles LLC, Pico Rivera, California
  - Pacific Clinical Research Medical Group, Riverside, California
  - California Neuropsychopharmacology Clinical Research Inst, San Diego, California
  - Stanford University, Stanford, California
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Fidelity Clinical Research, Lauderhill, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Center for Clinical Research, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Psychiatric Medicine Associates, Skokie, Illinois
  - Capital Clinical Research Associates, Rockville, Maryland
  - CNS Research Institute, Clementon, New Jersey
  - Behavioral Medical Research of Brooklyn, Brooklyn, New York
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Social Psychiatry Research Institute, New York, New York
  - Medical & Behavioral Health Research, New York, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Richard Weisler, MD and Associates, Raleigh, North Carolina
  - Piedmont Clinical Trials, Inc., Winston-Salem, North Carolina
  - Mood Disorders Program, Cleveland, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - Dubois Regional Medical Center - Behavioral Health Services, DuBois, Pennsylvania
  - Keystone Clinical Studies LLC, Norristown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Community Clinical Research, Austin, Texas
  - Claghorn-Lesem Research Clinic, LTD, Bellaire, Texas
  - University Hills Clinical Research, Irving, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington
- Bulgaria (5):
  - Call For Information, Burgas
  - Call For Information - Center Site #2, Plovdiv
  - Call For Information, Plovdiv
  - Call For Information - Center Site #2, Sofia
  - Call For Information, Sofia
- Hungary (2):
  - Call For Information, Budapest
  - Call For Information, Nagykálló
- Romania (4):
  - Call For Information, Bucharest
  - Call For Information - Center Site #2, Bucharest
  - Call For Information, Piteşti
  - Call For Information, Târgovişte

REFERENCES:
- [Derived] Calabrese JR, Ketter TA, Youakim JM, Tiller JM, Yang R, Frye MA. Adjunctive armodafinil for major depressive episodes associated with bipolar I disorder: a randomized, multicenter, double-blind, placebo-controlled, proof-of-concept study. J Clin Psychiatry. 2010 Oct;71(10):1363-70. doi: 10.4088/JCP.09m05900gry. Epub 2010 Jul 27. PMID 20673554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 centers in the US, Romania, Bulgaria, and Hungary. First participant enrolled: June 2007/ Last participant last visit: December 2008
Pre-assignment Details: The study consisted of a 1 to 2 week screening period, an 8 week double blind treatment period, and a 1 week follow up period.
Groups:
- Armodafinil 150 mg/Day: Armodafinil was titrated up to the target dosage of 150 mg/day (daily dose was administered each morning). Patients began taking blinded armodafinil at a dose of 50 mg/day (1 tablet) on the day following the baseline visit. Doses were increased by 50 mg/day (1 tablet) to a dose of 100 mg/day on Day 2 and 3, and then again by 50 mg /day on day 4 for a target dose of 150 mg/day. Following titration, patients continued taking 150 mg/day of armodafinil for the duration of the study. If a patient was unable to tolerate (recurrent or persistent adverse events) the study drug, 1 reduction in dosage (ie, minimum dosage 100 mg/day [2 tablets]) was allowed. The dosage could not be increased after it was decreased.
- Placebo: Placebo tablets matching the 50 mg armodafinil tablet were used in a manner identical to that of the armodafinil tablets. Study drug was titrated up to the target dosage of 3 tablets / day (daily dose was administered each morning). Patients began taking blinded study drug at a dose of 1 tablet daily on the day following the baseline visit. Doses were increased by 1 tablet to a dose of 2 tablets/day on Day 2 and 3, and then again by 1 tablet /day on day 4 for a target dose of 3 tablets/day. Following titration, patients continued taking 3 tablets/day of study drug for the duration of the study. If a patient was unable to tolerate (recurrent or persistent adverse events) the study drug, 1 reduction in dosage (ie, minimum dosage 2 tablets/day) was allowed. The dosage could not be increased after it was decreased.
Period: Overall Study
Arm/Group | Armodafinil 150 mg/Day | Placebo
Started | 128 (Two of these subjects were randomized but never received study medication.) | 129 (Four of these subjects were randomized but never received study medication.)
Completed | 89 | 90
Not Completed | 39 | 39
Not completed — Adverse Event | 16 | 11
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 4 | 6
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 10 | 7
Not completed — Withdrawal by Subject | 3 | 9
Not completed — Miscellaneous | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil 150 mg/Day | Placebo | Total
Number analyzed (Participants) | 128 | 129 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 128 | 129 | 257
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.6 (11.34) | 44.9 (11.53) | 43.7 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 76 | 140
  Male | 64 | 53 | 117
Region of Enrollment [Number; unit: participants]
  United States | 115 | 105 | 220
  Hungary | 0 | 2 | 2
  Romania | 5 | 7 | 12
  Bulgaria | 8 | 15 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change From Baseline to Endpoint (Week 8 or Last Observation After Baseline) in the 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30)
Description: The IDS C30 is a standardized 30 item, clinician rated scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data presented here summarizes the change from baseline to Endpoint (either week 8 or the last observation after baseline) in the total score of the IDS-C30.
Time Frame: Baseline and 8 weeks from start of study drug administration (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed with the IDS-C30 at both baseline and at least one time point after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 124 | 123
Units on a scale | -15.6 (1.32) | -12.5 (1.34)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Least square (LS) mean and standard error of the LS mean for each treatment group and the p-value for the treatment comparison is from an analysis of variance (ANOVA) with treatment ands concurrent treatment for bipolar disorders as factors. A significant treatment-by baseline interaction was observed in the total score that violates the assumption of parallelism on which an ANCOVA is based, so the data was analyzed using ANOVA without baseline as a covariate rather than ANCOVA; Test type: Superiority or Other; p = 0.0439, ANOVA

2. Secondary Outcome: The Mean Change From Baseline to Week 1 in the 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data presented here summarizes the change from baseline to Week 1 in the total score of the IDS-C30.
Time Frame: Baseline and 1 week following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed with the IDS-C30 at both baseline and at week 1 after start of study drug administration
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 120 | 118
Units on a scale | -6.5 (0.84) | -4.8 (0.85)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Least square (LS) mean and standard error of the LS mean for each treatment group and the p-value for the treatment comparison is from an ANCOVA with treatment and concurrent treatment for bipolar disorder as factors, and the baseline value as covariate; Test type: Superiority or Other; p = 0.0795, ANCOVA

3. Secondary Outcome: The Mean Change From Baseline to Week 2 in the 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data presented here summarizes the change from baseline to Week 2 in the total score of the IDS-C30.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed with the IDS-C30 at baseline and at 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 108 | 112
Units on a scale | -10.0 (1.04) | -7.3 (1.05)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0272, ANCOVA

4. Secondary Outcome: The Mean Change From Baseline to Week 3 in the 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data presented here summarizes the change from baseline to Week 3 in the total score of the IDS-C30.
Time Frame: Baseline and 3 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed with the IDS-C30 at baseline and at 3 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 102 | 100
Units on a scale | -13.1 (1.16) | -10.7 (1.20)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0802, ANCOVA

5. Secondary Outcome: The Mean Change From Baseline to Week 4 in the 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data presented here summarizes the change from baseline to Week 4 in the total score of the IDS-C30.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed with the IDS-C30 at baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 99 | 97
Units on a scale | -13.7 (1.19) | -12.1 (1.25)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2407, ANCOVA

6. Secondary Outcome: The Mean Change From Baseline to Week 6 in the 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data presented here summarizes the change from baseline to Week 6 in the total score of the IDS-C30.
Time Frame: Baseline and 6 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed with the IDS-C30 at baseline and at 6 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 92 | 92
Units on a scale | -16.7 (1.36) | -13.7 (1.40)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0502, ANCOVA

7. Secondary Outcome: The Mean Change From Baseline to Week 8 in the 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data presented here summarizes the change from baseline to Week 8 in the total score of the IDS-C30.
Time Frame: Baseline and 8 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed at baseline and at 8 weeks with the IDS-C30.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 89 | 90
Units on a scale | -17.8 (1.41) | -14.8 (1.45)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0612, ANCOVA

8. Secondary Outcome: Number of Patients Achieving Remission at Endpoint According to the 30-item Inventory of Depressive Symptomatology-Clinician-Rated (IDS-C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data here summarizes the number of subjects in each treatment group who achieved a remission (total score <=11).
Time Frame: Baseline, 4 and 8 weeks following start of study drug administration (or last observation after baseline)
Population: Full analysis set defined as subjects who had completed IDS-C30 at baseline and at least one observation after baseline
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 124 | 123
Participants
  Remission | 30 | 22
  No Remission | 94 | 101
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.1980, Cochran-Mantel-Haenszel — P-value is from a Cochran-Mantel-Haenzel chi-square test adjusted for concurrent treatment for bipolar disorder

9. Secondary Outcome: Number of Patients Achieving "Response" at Endpoint According to the 30-item Inventory of Depressive Symptomatology-Clinician-Rated (IDS-C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data here summarizes the number of subjects in each treatment group who achieved a "response" (> 50% decrease from baseline in total score).
Time Frame: Baseline, 4 and 8 weeks following start of study drug administration (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed by IDS-C30 at baseline, and at least one observation after baseline
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 124 | 123
Participants
  Response | 46 | 47
  No Response | 78 | 76
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.8960, Cochran-Mantel-Haenszel — P-value is from a Cochran-Mantel-Haenzel chi-square test adjusted for concurrent treatment for bipolar disorder

10. Secondary Outcome: Number of Patients Achieving "Sustained Remission" at Endpoint According to the 30-item Inventory of Depressive Symptomatology-Clinician-Rated (IDS-C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data here summarizes the number of subjects in each treatment group who achieved a "sustained remission" (total score <= 11 that persists over the four week period from Week 4 to Week 8).
Time Frame: Baseline, 4 and 8 weeks following start of study drug administration (or last observation after baseline)
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 124 | 123
Participants
  Sustained Remission | 13 | 8
  No Sustained Remission | 111 | 115
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.2575, Cochran-Mantel-Haenszel — P-value is from a Cochran-Mantel-Haenzel chi-square test adjusted for concurrent treatment for bipolar disorder

11. Secondary Outcome: Number of Patients Achieving "Sustained Response" at Endpoint According to the 30-item Inventory of Depressive Symptomatology-Clinician-Rated (IDS-C30)
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. The data here summarizes the number of subjects in each treatment group who achieved a "sustained response" (> 50% decrease from baseline in total score that persisted over the four week period between Week 4 and Week 8).
Time Frame: Baseline, 4 and 8 weeks following start of study drug administration (or last observation after baseline)
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 124 | 123
Participants
  Sustained Response | 23 | 17
  No Sustained Response | 101 | 106
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.3129, Cochran-Mantel-Haenszel — P-value is from a Cochran-Mantel-Haenzel chi-square test adjusted for concurrent treatment for bipolar disorder

12. Secondary Outcome: Change From Baseline to Endpoint (Week 8 or Last Observation After Baseline) on 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30) Combination of Items 1-3
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. Items 1 - 3 assess sleep onset insomnia, mid-nocturnal insomnia, and early morning insomnia respectively each on a 0 - 3 scale. The data presented here summarizes the change from baseline to Endpoint in the combined score of these three items assessing insomnia.
Time Frame: Baseline and 8 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects who were assessed by IDS-C30 at baseline and at least one observation after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 124 | 123
Units on a scale | -1.6 (0.24) | -1.2 (0.25)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1565, ANCOVA

13. Secondary Outcome: Change From Baseline to Week 4 on 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30) Combination of Items 1-3
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. Items 1 - 3 assess sleep onset insomnia, mid-nocturnal insomnia, and early morning insomnia respectively each on a 0 - 3 scale. The data presented here summarizes the change from baseline to week 4 in the combined score of these three items assessing insomnia.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed by IDS C30 at baseline and Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 99 | 97
Units on a scale | -1.2 (0.26) | -1.1 (0.27)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6737, ANCOVA

14. Secondary Outcome: Change From Baseline to Week 8 on 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30) Combination of Items 1-3
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. Items 1 - 3 assess sleep onset insomnia, mid-nocturnal insomnia, and early morning insomnia respectively each on a 0 - 3 scale. The data presented here summarizes the change from baseline to week 8 in the combined score of these three items assessing insomnia.
Time Frame: Baseline and 8 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed with IDS-C30 at baseline and at week 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 89 | 90
Units on a scale | -2.0 (0.28) | -1.6 (0.28)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2249, ANCOVA

15. Secondary Outcome: Change From Baseline to Endpoint (Week 8 or Last Observation After Baseline) on 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30) - Item 4
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. Item 4 assesses hypersomnia on a scale from 0 (sleeps no longer than 7-8 hours a night) to 3 (sleeps longer than 12 hours in 24 hour period). The data presented here summarizes the change from baseline to Endpoint in the score of Item 4 assessing hypersomnia.
Time Frame: Baseline and 8 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects assessed with IDS-C30 at baseline and at least one observation after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 124 | 123
Units on a scale | -0.4 (0.06) | -0.2 (0.07)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0862, ANCOVA

16. Secondary Outcome: Change From Baseline to Week 4 on 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30) - Item 4
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. Item 4 assesses hypersomnia on a scale from 0 (sleeps no longer than 7-8 hours a night) to 3 (sleeps longer than 12 hours in 24 hour period). The data presented here summarizes the change from baseline to week 4 in the score of Item 4 assessing hypersomnia.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects assessed with IDS-C30 at baseline and at week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 99 | 97
Units on a scale | -0.2 (0.07) | -0.2 (0.07)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9281, ANCOVA

17. Secondary Outcome: Change From Baseline to Week 8 on 30 Item Inventory of Depressive Symptomatology Clinician Rated (IDS C30) - Item 4
Description: The IDS C30 is a standardized 30 item, clinician rated, scale to assess the severity of a patient's depressive symptoms. The scale uses the 9 symptom domains of the DSM-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression. Item 4 assesses hypersomnia on a scale from 0 (sleeps no longer than 7-8 hours a night) to 3 (sleeps longer than 12 hours in 24 hour period). The data presented here summarizes the change from baseline to week 8 in the score of Item 4 assessing hypersomnia.
Time Frame: Baseline and 8 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed with IDS-C30 at baseline and at week 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 89 | 90
Units on a scale | -0.3 (0.08) | -0.2 (0.08)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4428, ANCOVA

18. Secondary Outcome: Change From Baseline to Endpoint (Week 8 or Last Observation After Baseline) in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item scale to evaluate the overall severity of a patient's depressive symptoms, that is completed by the physician. The rating scale makes use of both observational clues as to the subject's level of depression (eg. apparent sadness) and verbal indicators of depression expressed by the patient. Each of the 10 items is graded on a 6-point scale with anchors at 2 point intervals. Total scores range from 0 to 60, with the higher number indicating more severe symptoms of depression. Here we present data summarizing the change in MADRS from Baseline to Endpoint.
Time Frame: Baseline and Endpoint (8 weeks following the start of study drug administration or last observation after baseline)
Population: Full analysis set defined as subjects who had both a baseline observation and at least one observation after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 118 | 116
Units on a scale | -12.3 (1.10) | -10.2 (1.12)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0965, ANCOVA

19. Secondary Outcome: Change From Baseline to Week 4 in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item scale to evaluate the overall severity of a patient's depressive symptoms, that is completed by the physician. The rating scale makes use of both observational clues as to the subject's level of depression (eg. apparent sadness) and verbal indicators of depression expressed by the patient. Each of the 10 items is graded on a 6-point scale with anchors at 2 point intervals. Total scores range from 0 to 60, with the higher number indicating more severe symptoms of depression. Here we present data summarizing the difference in MADRS score from Baseline to Week 4.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed by MADRS at both baseline and at Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 99 | 97
Units on a scale | -9.6 (1.03) | -8.9 (1.08)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5389, ANCOVA

20. Secondary Outcome: Change From Baseline to Week 8 in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item scale to evaluate the overall severity of a patient's depressive symptoms, that is completed by the physician. The rating scale makes use of both observational clues as to the subject's level of depression (eg. apparent sadness) and verbal indicators of depression expressed by the patient. Each of the 10 items is graded on a 6-point scale with anchors at 2 point intervals. Total scores range from 0 to 60, with the higher number indicating more severe symptoms of depression. Here we present data summarizing the difference in MADRS score from Baseline to Week 8.
Time Frame: Baseline and 8 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed by MADRS at both baseline and at Week 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 89 | 90
Units on a scale | -13.4 (1.20) | -11.0 (1.24)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0793, ANCOVA

21. Secondary Outcome: Change From Baseline to Endpoint (Week 8 or Last Observation After Baseline) in the Quick Inventory of Depressive Symptomatology - 16 Items (QIDS-SR16)
Description: The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the patient at each visit. It is a shorter version of the IDS-C30 that is completed by the patient rather than the examiner. The total score ranges from 0 to 27 (higher score signifies more severe depression) and is obtained by adding the scores for each of the 9 depression symptom domains of the DSM IV. The data presented here summarizes the change in QIDS-SR16 from Baseline to Endpoint (Week 8 or last observation after baseline).
Time Frame: Baseline and 8 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects who completed the QIDS-SR16 at baseline and at least one observation after baseline.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 124 | 123
Units on a scale | -7.0 (0.55) | -6.5 (0.56)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3814, ANCOVA

22. Secondary Outcome: Change From Baseline to Week 1 in the Quick Inventory of Depressive Symptomatology - 16 Items (QIDS-SR16)
Description: The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the patient at each visit. It is a shorter version of the IDS-C30 that is completed by the patient rather than the examiner. The total score ranges from 0 to 27 (higher score signifies more severe depression) and is obtained by adding the scores for each of the 9 depression symptom domains of the DSM IV. The data presented here summarizes the change in QIDS-SR16 from Baseline to Week 1
Time Frame: Baseline and 1 week following the start of study drug administration
Population: Full analysis set defined as subjects who completed the QIDS-SR16 at baseline and at 1 week
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 120 | 118
Units on a scale | -3.5 (0.42) | -3.7 (0.43)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8099, ANCOVA

23. Secondary Outcome: Change From Baseline to Week 2 in the Quick Inventory of Depressive Symptomatology - 16 Items (QIDS-SR16)
Description: The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the patient at each visit. It is a shorter version of the IDS-C30 that is completed by the patient rather than the examiner. The total score ranges from 0 to 27 (higher score signifies more severe depression) and is obtained by adding the scores for each of the 9 depression symptom domains of the DSM IV. The data presented here summarizes the change in QIDS-SR16 from Baseline to Week 2
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the QIDS-SR16 at baseline and at 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 108 | 113
Units on a scale | -5.0 (0.44) | -4.1 (0.44)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0968, ANCOVA

24. Secondary Outcome: Change From Baseline to Week 3 in the Quick Inventory of Depressive Symptomatology - 16 Items (QIDS-SR16)
Description: The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the patient at each visit. It is a shorter version of the IDS-C30 that is completed by the patient rather than the examiner. The total score ranges from 0 to 27 (higher score signifies more severe depression) and is obtained by adding the scores for each of the 9 depression symptom domains of the DSM IV. The data presented here summarizes the change in QIDS-SR16 from Baseline to Week 3.
Time Frame: Baseline and 3 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the QIDS-SR16 at baseline and at week 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 102 | 101
Units on a scale | -5.8 (0.52) | -5.0 (0.54)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1605, ANCOVA

25. Secondary Outcome: Change From Baseline to Week 4 in the Quick Inventory of Depressive Symptomatology - 16 Items (QIDS-SR16)
Description: The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the patient at each visit. It is a shorter version of the IDS-C30 that is completed by the patient rather than the examiner. The total score ranges from 0 to 27 (higher score signifies more severe depression) and is obtained by adding the scores for each of the 9 depression symptom domains of the DSM IV. The data presented here summarizes the change in QIDS-SR16 from Baseline to Week 4.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the QIDS-SR16 at baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 99 | 97
Units on a scale | -6.4 (0.53) | -5.6 (0.56)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1869, ANCOVA

26. Secondary Outcome: Change From Baseline to Week 6 in the Quick Inventory of Depressive Symptomatology - 16 Items (QIDS-SR16)
Description: The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the patient at each visit. It is a shorter version of the IDS-C30 that is completed by the patient rather than the examiner. The total score ranges from 0 to 27 (higher score signifies more severe depression) and is obtained by adding the scores for each of the 9 depression symptom domains of the DSM IV. The data presented here summarizes the change in QIDS-SR16 from Baseline to Week 6.
Time Frame: Baseline and 6 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the QIDS-SR16 at baseline and at 6 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 92 | 92
Units on a scale | -7.8 (0.58) | -6.7 (0.60)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0817, ANCOVA

27. Secondary Outcome: Change From Baseline to Week 8 in the Quick Inventory of Depressive Symptomatology - 16 Items (QIDS-SR16)
Description: The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the patient at each visit. It is a shorter version of the IDS-C30 that is completed by the patient rather than the examiner. The total score ranges from 0 to 27 (higher score signifies more severe depression) and is obtained by adding the scores for each of the 9 depression symptom domains of the DSM IV. The data presented here summarizes the change in QIDS-SR16 from Baseline to Week 8.
Time Frame: Baseline and 8 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the QIDS-SR16 at baseline and at 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 89 | 90
Units on a scale | -8.2 (0.58) | -7.6 (0.60)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3712, ANCOVA

28. Secondary Outcome: Change From Baseline to Endpoint (Week 8 or Last Observation After Baseline) in the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF)
Description: The Q-LES-Q-SF is an instrument designed to measure general activities of daily living. It is a patient-rated quality of life questionnaire and consists of 16 items, but only the first 14 are included in the total score. Each item is rated by the patient on a scale from 1 - 5 (1=very poor, 2=poor, 3=fair, 4=good, and 5=very good). The minimum score is 14 and the maximum score is 70, with lower scores indicating poorer quality of life. The data presented here summarizes the change in score from baseline to endpoint (8 weeks or last observation after baseline).
Time Frame: Baseline and 8 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects who completed the questionnaire at baseline and at any appropriate time point after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 115 | 112
Units on a scale | 8.2 (1.12) | 7.4 (1.16)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5427, ANCOVA

29. Secondary Outcome: Change From Baseline to Week 4 in the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF)
Description: The Q-LES-Q-SF is an instrument designed to measure general activities of daily living. It is a patient-rated quality of life questionnaire and consists of 16 items, but only the first 14 are included in the total score. Each item is rated by the patient on a scale from 1 - 5 (1=very poor, 2=poor, 3=fair, 4=good, and 5=very good). The minimum score is 14 and the maximum score is 70, with lower scores indicating poorer quality of life. The data presented here summarizes the change in score from baseline to 4 weeks.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the questionnaire at baseline and at 4 weeks.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 95 | 95
Units on a scale | 5.9 (1.16) | 4.6 (1.22)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3463, ANCOVA

30. Secondary Outcome: Change From Baseline to Week 8 in the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF)
Description: The Q-LES-Q-SF is an instrument designed to measure general activities of daily living. It is a patient-rated quality of life questionnaire and consists of 16 items, but only the first 14 are included in the total score. Each item is rated by the patient on a scale from 1 - 5 (1=very poor, 2=poor, 3=fair, 4=good, and 5=very good). The minimum score is 14 and the maximum score is 70, with lower scores indicating poorer quality of life. The data presented here summarizes the change in score from baseline to 8 weeks.
Time Frame: Baseline and 8 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed questionnaire at baseline and at 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 85 | 86
Units on a scale | 10.1 (1.29) | 8.5 (1.34)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2730, ANCOVA

31. Secondary Outcome: Change From Baseline to Endpoint (8 Weeks or Last Observation After Baseline) in Hamilton Anxiety Scale (HAM-A) Total Score
Description: The HAM-A is a clinician-rated 14 item scale that provides an overall measure of global anxiety, including psychic (mental agitation and psychological distress) and somatic (physical complaints related to anxiety) symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0 - 56, where less than 17 indicates mild anxiety, 18 - 24 mild to moderate anxiety, 25-30 moderate to severe, >30 very severe. The data presented here summarizes the change in HAM-A score from Baseline to Endpoint (8 weeks or last observation after baseline).
Time Frame: baseline and 8 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects who completed the HAM-A at baseline and at least once after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 117 | 116
Units on a scale | -4.1 (0.60) | -3.9 (0.61)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7791, ANCOVA

32. Secondary Outcome: Change From Baseline to 4 Weeks in the Hamilton Anxiety Scale (HAM A) Total Score
Description: The HAM-A is a clinician-rated 14 item scale that provides an overall measure of global anxiety, including psychic (mental agitation and psychological distress) and somatic (physical complaints related to anxiety) symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0 - 56, where less than 17 indicates mild anxiety, 18 - 24 mild to moderate anxiety and 25-30 moderate to severe. The data presented here summarizes the change in HAM-A score from Baseline to 4 Weeks
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the HAM-A at baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 99 | 97
Units on a scale | -3.6 (0.58) | -3.5 (0.60)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9007, ANCOVA

33. Secondary Outcome: Change From Baseline to 8 Weeks in the Hamilton Anxiety Scale (HAM A) Total Score
Description: The HAM-A is a clinician-rated 14 item scale that provides an overall measure of global anxiety, including psychic (mental agitation and psychological distress) and somatic (physical complaints related to anxiety) symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0 - 56, where less than 17 indicates mild anxiety, 18 - 24 mild to moderate anxiety and 25-30 moderate to severe. The data presented here summarizes the change in HAM-A score from Baseline to 8 Weeks
Time Frame: Baseline and 8 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the HAM-A at baseline and at 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 89 | 90
Units on a scale | -4.7 (0.68) | -4.4 (0.70)
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6431, ANCOVA

34. Secondary Outcome: The Number of Responders According to the Clinical Global Impression of Change - Bipolar Version (CGI BP) Measure of Depression at Endpoint (Week 8 or Last Observation After Baseline)
Description: CGI-BP is a standardized, clinician-rated assessment which allows the clinician to rate the bipolar illness at various time points compared with baseline. At Screening and Baseline visits the physician rated the severity of the illness using 7 categories (1=normal through 7=very severely ill). At subsequent visits the clinician assessed the change in severity of the condition using 7 categories (1=very much improved through 7=very much worse). Subjects were considered responders if they had a rating of "much improved" or "very much improved". The number of responders at Endpoint are presented.
Time Frame: Baseline and 8 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects assessed by CGI-BP at Baseline and at least one observation after Baseline.
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 124 | 122
Participants
  Responder | 64 | 60
  Non Responder | 60 | 62
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.6631, Cochran-Mantel-Haenszel; Adjusted for concurrent treatment for bipolar disorder

35. Secondary Outcome: The Number of Responders According to the Clinical Global Impression of Change - Bipolar Version (CGI BP) Measure of Depression at Week 1
Description: CGI-BP is a standardized, clinician-rated assessment which allows the clinician to rate the bipolar illness at various time points compared with baseline. At Screening and Baseline visits the physician rated the severity of the illness using 7 categories (1=normal through 7=very severely ill). At subsequent visits the clinician assessed the change in severity of the condition using 7 categories (1=very much improved through 7=very much worse). Subjects were considered responders if they had a rating of "much improved" or "very much improved". The number of responders at Week 1 are presented.
Time Frame: Baseline and 1 week following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed by CGI-BP at Baseline and Week 1
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 119 | 117
Participants
  Responder | 12 | 12
  Non Responder | 107 | 105
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.9768, Cochran-Mantel-Haenszel; Adjusted for concurrent treatment for bipolar disorder

36. Secondary Outcome: The Number of Responders According to the Clinical Global Impression of Change - Bipolar Version (CGI BP) Measure of Depression at Week 2
Description: CGI-BP is a standardized, clinician-rated assessment which allows the clinician to rate the bipolar illness at various time points compared with baseline. At Screening and Baseline visits the physician rated the severity of the illness using 7 categories (1=normal through 7=very severely ill). At subsequent visits the clinician assessed the change in severity of the condition using 7 categories (1=very much improved through 7=very much worse). Subjects were considered responders if they had a rating of "much improved" or "very much improved". The number of responders at Week 2 are presented.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed by CGI-BP at baseline and week 2
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 108 | 110
Participants
  Responder | 25 | 26
  Non Responder | 83 | 84
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.9873, Cochran-Mantel-Haenszel; Adjusted for concurrent treatment fro bipolar disorder

37. Secondary Outcome: The Number of Responders According to the Clinical Global Impression of Change - Bipolar Version (CGI BP) Measure of Depression at Week 3
Description: CGI-BP is a standardized, clinician-rated assessment which allows the clinician to rate the bipolar illness at various time points compared with baseline. At Screening and Baseline visits the physician rated the severity of the illness using 7 categories (1=normal through 7=very severely ill). At subsequent visits the clinician assessed the change in severity of the condition using 7 categories (1=very much improved through 7=very much worse). Subjects were considered responders if they had a rating of "much improved" or "very much improved". The number of responders at Week 3 are presented.
Time Frame: Baseline and 3 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed by CGI-BP at baseline and at 3 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 102 | 100
Participants
  Responder | 38 | 32
  Non Responder | 64 | 68
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.4567, Cochran-Mantel-Haenszel; Adjusted for concurrent treatment for bipolar disorder

38. Secondary Outcome: The Number of Responders According to the Clinical Global Impression of Change - Bipolar Version (CGI BP) Measure of Depression at Week 4
Description: CGI-BP is a standardized, clinician-rated assessment which allows the clinician to rate the bipolar illness at various time points compared with baseline. At Screening and Baseline visits the physician rated the severity of the illness using 7 categories (1=normal through 7=very severely ill). At subsequent visits the clinician assessed the change in severity of the condition using 7 categories (1=very much improved through 7=very much worse). Subjects were considered responders if they had a rating of "much improved" or "very much improved". The number of responders at Week 4 are presented.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed with CGI-BP at baseline and at 4 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 99 | 97
Participants
  Responder | 46 | 42
  Non Responder | 53 | 55
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.6475, Cochran-Mantel-Haenszel; Adjusted for concurrent treatment for bipolar disorder

39. Secondary Outcome: The Number of Responders According to the Clinical Global Impression of Change - Bipolar Version (CGI BP) Measure of Depression at Week 6
Description: CGI-BP is a standardized, clinician-rated assessment which allows the clinician to rate the bipolar illness at various time points compared with baseline. At Screening and Baseline visits the physician rated the severity of the illness using 7 categories (1=normal through 7=very severely ill). At subsequent visits the clinician assessed the change in severity of the condition using 7 categories (1=very much improved through 7=very much worse). Subjects were considered responders if they had a rating of "much improved" or "very much improved". The number of responders at Week 6 are presented.
Time Frame: Baseline and 6 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed by CGI-BP at baseline and at Week 6
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 92 | 92
Participants
  Responder | 47 | 43
  Non Responder | 45 | 49
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.5066, Cochran-Mantel-Haenszel; Adjusted for concurrent treatment for bipolar disorder

40. Secondary Outcome: The Number of Responders According to the Clinical Global Impression of Change - Bipolar Version (CGI BP) Measure of Depression at Week 8
Description: CGI-BP is a standardized, clinician-rated assessment which allows the clinician to rate the bipolar illness at various time points compared with baseline. At Screening and Baseline visits the physician rated the severity of the illness using 7 categories (1=normal through 7=very severely ill). At subsequent visits the clinician assessed the change in severity of the condition using 7 categories (1=very much improved through 7=very much worse). Subjects were considered responders if they had a rating of "much improved" or "very much improved". The number of responders at Week 8 are presented.
Time Frame: Baseline and 8 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who were assessed with CGI-BP at baseline and at week 8
Measure: Number; unit: Participants
Arm/Group | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 89 | 88
Participants
  Responder | 52 | 47
  Non Responder | 37 | 41
Statistical Analysis 1: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.4438, Cochran-Mantel-Haenszel; Adjusted for concurrent treatment for bipolar disorder

ADVERSE EVENTS:
Arm/Group | Armodafinil 150 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 3/126 | 3/125
Other Adverse Events (participants affected / at risk) | 56/126 | 54/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil 150 mg/Day (N=126) | Placebo (N=125)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 2 (2)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 150 mg/Day (N=126) | Placebo (N=125)
Diarrhoea (Gastrointestinal disorders) | 12 | 8
Nausea (Gastrointestinal disorders) | 9 | 6
Dry Mouth (Gastrointestinal disorders) | 8 | 5
Vomiting (Gastrointestinal disorders) | 5 | 4
Toothache (Gastrointestinal disorders) | 1 | 5
Fatigue (General disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 9
Nasopharyngitis (Infections and infestations) | 2 | 4
Weight increased (Investigations) | 1 | 6
Headache (Nervous system disorders) | 14 | 12
Somnolence (Nervous system disorders) | 6 | 2
Tremor (Nervous system disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 13 | 10
Restlessness (Psychiatric disorders) | 7 | 1
Anxiety (Psychiatric disorders) | 5 | 2
Mania (Psychiatric disorders) | 1 | 4
Initial insomnia (Psychiatric disorders) | 0 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days